CLINICAL TRIAL: NCT05250323
Title: Energy Balance in Huntington's Disease. A Multidisciplinary Study Approach for a Complex Problem (BEHD-EM)
Acronym: BEHD-EM
Status: Completed | Type: Observational
Sponsor: Hospital Universitario de Burgos (Other)
Collaborators: La Caixa Foundation (Other); Universidad Isabel I (Unknown)
Responsible Party: Principal Investigator, Esther Cubo, Dr. Neurology, Hospital Universitario de Burgos
Other Study IDs: CEIM-2429
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Huntington Disease
Keywords: energy expenditure; physical activity; nutrition; wereables; daily life activity
MeSH Terms: conditions — Huntington Disease; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with genetic confirmation of Huntington's disease, symptomatic (motor manifestations with a score greater than 4 on the Unified HD scale), who can walk with minimal support, without sensory deficits or other systemic diseases an Investigator judgment that may interfere with the execution of the study, coming from the Enroll study.
  Interventions: Other: observational tests in face-to-face visit
- Control: Age, gender-matched non-gene carriers family relatives
  Interventions: Other: observational tests in face-to-face visit

INTERVENTIONS:
Other: observational tests in face-to-face visit — All necessary evaluations will be carried out for data collection. Also, that same day, the investigators will give the device to participants for the 7-day home assessment

SUMMARY:
The study was conducted at the University Isabel I, Burgos in collaboration with the Hospital Universitario Burgos, Spain, through the creation of a multidisciplinary research team including graduates in physical activity and sports sciences, dietitians-nutritionists, neurologists and occupational therapists. To carry out this study: 1) the investigators used new technologies, specifically, small wearable or wearable devices available to the population. These devices measure their daily behaviour and estimate aspects such as energy expenditure, validated both in healthy participants and in participants with neurodegenerative diseases such as Parkinson's disease, but not in HD; 2) the investigators included a consecutive sample of patients with HD ; 3) the investigators performed the experimental study at the the laboratory for Exercise Physiology, Health and Quality of Life at the Isabel I University.

The hypothesis proposed by this study are the following: 1) Patients with HD who present an adequate energy balance caused by healthier lifestyles (active lifestyles and healthy eating) will present a better functional capacity, quality of life and therefore both less dependency; 2) HD patients with a balanced energy balance maintain adequate body composition (muscle, fat); 3) Adequate body composition is associated with better functional capacity in HD patients.

DETAILED DESCRIPTION:
In the last decade, numerous studies have been published showing how epigenetic (environmental) factors can modify the clinical manifestations of diseases of genetic origin. Specifically, epidemiological studies have observed that physical exercise delays the onset and slows down the progression of neurodegenerative diseases (dementia, Parkinson's disease, HD), by producing, between the different mechanisms, greater plasticity of the different neuronal circuits. Another environmental factor such as nutrition has also been highlighted by numerous authors, highlighting the role of the Mediterranean diet in delaying the onset, especially in Parkinson's disease, as the phenolic components of olive oil produce an inhibition of the Pathological aggregation of modified alpha synuclein. On the contrary, it has been seen that an energy deficit at the cellular level accelerates the neurodegeneration process, shortening survival in different animal models.

To maintain an adequate energy balance, it is required that the energy expenditure produced by physical activity (GAF), plus the expenditure produced by the maintenance of the different organs: energy expenditure at rest (GAR) and thermogenesis, is similar to the input of energy produced by the oxidation of macronutrients from food intake. In HD, it is believed that this energy balance is not adequate, either due to the decrease in food intake (very frequent when there are swallowing problems), and the decrease in physical activity produced by alterations in mobility, or by structural damage (hypothalamic, mitochondrial) produced by the neurodegeneration process per se. When the energy balance is negative (energy expenditure> caloric intake), due to a decrease in intake or due to sustained involuntary physical activity (chorea), it can lead to the use of other energy substrates such as adipose tissue and muscle, triggering sarcopenia, cachexia, and ultimately, accelerating the neurodegeneration process. Weight loss and a low body mass index (BMI) in patients with neurodegenerative diseases lead to a greater development of neurological symptoms, while a high food intake has been associated with a more rapid progression in the symptoms of these patients. For all these reasons, it seems that nutrition plays a determining role, the dietary and nutritional analysis being fundamental.

To date, there are very few studies on energy balance in neurodegenerative diseases, addressing it from a comprehensive point of view and analysing each of its contributing components (energy expenditure-caloric intake). A better knowledge of the energy balance in HD may lead to the development of non-pharmacological, easily accessible and cost-effective therapeutic strategies such as lifestyle modifications, through adequate physical activity and nutritional intake.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old
* Genetic confirmation of Huntington's disease
* Symptomatic (motor manifestations with a score greater than 4 on the Unified HD scale)
* Walk with minimal support
* Participate in Enroll study
* Non-gene carriers, family relatives

Exclusion Criteria:

* Sensory deficits or other systemic diseases which according to the Investigator judgment may interfere with the execution of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with Huntington's disease and non-gene family relatives
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Measurement of energy expenditure at rest | 10 minutes
  by indirect calorimetry recording respiratory exchange (Medisoft Ergocard, Medisoft Group, Sorinnes, Belgium)
Measurement of energy expenditure due to physical activity | 45 minutes
  using a wearable device (Fitbit Charge), which allows quantification in a valid and reliable way, in patients with HD
Determination of caloric intake | 30 minutes
  by registering eating habits (SUN food frequency questionnaire and a 3-day food diary)
Bone densitometry (DXA) | 10 minutes
  Determination of body composition

SECONDARY OUTCOMES:
Validation of the wearable comparing the results with a gold standard | 45 minutes
  using indirect calorimetry and accelerometery (ActiGraph wGT3X-BT) during activities of various kinds and intensity (walking at different speeds and slopes) on a treadmill (h / p / cosmos pulsar, h / p / cosmos sports and medical GMBH, Nussdorf-Traunstein, Germany) and activities of daily living together with pedalling on a cycle ergometer
Determination of the incidence of thermogenesis on energy expenditure and on the appearance of fatigue | 2 hours
  by recording the central and peripheral temperature (VitalSense, Phillips Respironics, Bend, OR, USA).
Determination of lifestyle and weekly energy expenditure | 7 days
  for this the participants will wear the device for 7 consecutive days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No